CLINICAL TRIAL: NCT01305109
Title: A Phase III, Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Protective Efficacy of Three Doses of Oral Rotavirus Vaccine (ORV) 116E, Against Severe Rotavirus Gastroenteritis in Infants
Brief Title: A Phase III Clinical Trial to Evaluate the Protective Efficacy of Three Doses of Oral Rotavirus Vaccine (ORV) 116E
Acronym: ROTAVAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bharat Biotech International Limited (Industry)
Collaborators: Ministry of Science and Technology, India (Other Government); PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBIL/ROTA/021; Clinical Trials Registry-India (Registry Identifier: CTRI/2010/091/000102)
Record Dates: First submitted 2011-02-18; First posted 2011-02-28 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Viral Gastroenteritis Due to Rotavirus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Rotavirus Vaccine 116E (ORV 116E) (Experimental): Oral Rotavirus Vaccine 116E (ORV 116E), 10^5.0 FFU of Bharat Biotech International Limited, 3 doses of 0.5 mL at 4 week intervals
  Interventions: Biological: ORV 116E
- Placebo (Placebo Comparator): 3 doses of 0.5 mL at 4 week intervals
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ORV 116E — Oral Rotavirus Vaccine 116E (ORV 116E), 10^5.0 FFU of Bharat Biotech International Limited, 3 doses of 0.5mL at 4 week intervals
  Other Names: ROTAVAC
  Arms: Oral Rotavirus Vaccine 116E (ORV 116E)
Biological: Placebo — 3 doses of 0.5 mL at 4 week intervals
  Arms: Placebo

SUMMARY:
The trial is a phase III randomized, double-blind, placebo-controlled trial with the primary objective of evaluating the efficacy of three doses of ORV 116E, 10^5.0 FFU, against severe rotavirus gastroenteritis, in comparison with a placebo in India.

DETAILED DESCRIPTION:
The trial is a phase III randomized, double-blind, placebo-controlled trial with the primary objective of evaluating the efficacy of three doses of ORV 116E, 10^5.0 FFU, against severe rotavirus gastroenteritis, in comparison with a placebo in India. The clinical trial is not a global trial. Three administrations of ORV 116E will be co-administered with childhood vaccines (which will include vaccines against diphtheria, pertussis, tetanus, Haemophilus influenzae B and Hepatitis B and OPV) at 6 to 7 weeks, greater than or equal to 10 weeks and greater than or equal to 14 weeks of age. 6800 subjects will be enrolled in three sites - Delhi, Pune (Maharashtra) and Vellore (Tamil Nadu) and followed up till the age of 2 years (24 months + up to 14 days). Multiple trial sites are included to ensure greater demographic distribution to obtain evidence of cross immunity and quicker recruitment of the necessary number of subjects. The subjects to be included from these sites would be representative of the population of India.

The protocol has been reviewed by the institutional review boards of the Society for Applied Studies (New Delhi), KEM Hospital Research Centre (Pune), Christian Medical College (Vellore). Ethics clearance has also been obtained from the Department of Biotechnology, Government of India and Western Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* At least one parent(s) or legally acceptable representative's consent for participation and are able to understand study procedures
* Subjects aged 6 to 7 weeks at recruitment
* No plans to move in the next 24 months

Exclusion Criteria:

* Administration of rotavirus vaccine in the past
* Presence of any illness requiring hospital referral (temporary exclusion)
* Known case of immunodeficiency disease, known HIV positive
* Known case of chronic gastroenteritis disease
* Any other conditions which in the judgment of the investigator warrant exclusion (e.g. no exclusion criteria but seems "ill", investigators suspects neglect)
* Diarrhea on the day of enrollment (temporary exclusion)

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6800 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus in all subjects from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days.

SECONDARY OUTCOMES:
Efficacy against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus | Up to 1 year of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus occurring at least 14 days following the third dose till the age of 12 months + up to 14 days
Efficacy against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus | From the age of 12 months till the age of 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo for severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus occurring from the age of 12 months till the age of 2 years (24 months) + up to 14 days
Efficacy against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus in intent-to-treat population | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo against severe rotavirus gastroenteritis (>=11 on the 20 point Vesikari scoring scale) caused by non vaccine rotavirus in the intent-to-treat population till the age of 2 years (24 months) + up to 14 days.
Efficacy against any severity of gastroenteritis caused by a non vaccine rotavirus | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo for any severity of gastroenteritis caused by non vaccine rotavirus from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy against any severity of gastroenteritis irrespective of etiology | Up to 2 years of Age
  Efficacy of ORV 116E will be assessed in comparison to a placebo for any severity of gastroenteritis irrespective of etiology from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy against severe (>=11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo for severe (≥11 on the 20 point Vesikari scoring scale) gastroenteritis irrespective of etiology from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy to prevent hospitalization and/or supervised rehydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for gastroenteritis caused by non vaccine rotavirus | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for gastroenteritis caused by non vaccine rotavirus from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy to prevent hospitalization and/or supervised rehydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for gastroenteritis of any etiology | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for gastroenteritis of any etiology from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for severe gastroenteritis caused by non vaccine rotavirus | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for severe gastroenteritis caused by non vaccine rotavirus from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for severe gastroenteritis of any etiology | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to a placebo to prevent hospitalization and/or supervised re-hydration therapy (equivalent to WHO plan B or C) in a treatment facility/hospital for severe gastroenteritis of any etiology from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Efficacy against very severe rotavirus gastroenteritis (≥16 on the 20-point Vesikari scoring system) caused by non vaccine rotavirus | Up to 2 years of age
  Efficacy of ORV 116E will be assessed in comparison to placebo against very severe rotavirus gastroenteritis (≥16 on the 20-point Vesikari scoring system) caused by non vaccine rotavirus from 14 days following the 3rd dose till the age of 2 years (24 months) + up to 14 days
Safety of ORV 116E for immediate adverse events and serious adverse events in comparison to a placebo | Up to 2 years of age
  Safety of ORV 116E for immediate adverse events and serious adverse events in comparison to a placebo will be assessed in all the subjects, from day of 1st dose till the age of 2 years (24 months) + up to 14 days.
Safety of ORV 116E for adverse events in a subset | 2 weeks period following each administration
  Safety of ORV 116E for adverse events assessed daily in the 2 week period following each dose in comparison to a placebo in first one third of the enrolled subjects in all the three sites
Safety of ORV 116E for intussusception events | Up to 2 years of age
  Safety of ORV 116E for intussusception events in comparison to a placebo will be assessed in all subjects, from day of 1st dose till the age of 2 years (24 months) + up to 14 days
Immunogenicity rates to three doses of the ORV 116E and vaccine virus shedding rates after each of the three doses of the ORV 116E in a subset | 28 days after administration of third dose
  Immunogenicity rates to three doses of the ORV 116E and vaccine virus shedding rates after each of the three doses of the ORV 116E in comparison to a placebo will be ascertained in approximately 150 subjects at each site.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Temsunaro R Chandola, MD, MSc, Principal Investigator — Centre for Health Research and Development, Society for Applied Studies; Gagandeep Kang, MDFRCPathPhD, Principal Investigator — Christian Medical College, Vellore, India; Ashish Bavdekar, MD,DCH,DNB, Principal Investigator — Shirdi Sai Baba Rural Hospital, KEM Hospital Research Centre,Vadu Rural Health
Locations (3):
- India (3):
  - Shirdi Sai Baba Rural Hospital, KEM Hospital Research Centre,Vadu Rural Health, Pune, Maharashtra
  - Centre for Health Research and Development, Society for Applied Studies, New Delhi, New Delhi
  - Christian Medical College, Vellore

REFERENCES:
- [Derived] Bhandari N, Rongsen-Chandola T, Bavdekar A, John J, Antony K, Taneja S, Goyal N, Kawade A, Kang G, Rathore SS, Juvekar S, Muliyil J, Arya A, Shaikh H, Abraham V, Vrati S, Proschan M, Kohberger R, Thiry G, Glass R, Greenberg HB, Curlin G, Mohan K, Harshavardhan GV, Prasad S, Rao TS, Boslego J, Bhan MK; India Rotavirus Vaccine Group. Efficacy of a monovalent human-bovine (116E) rotavirus vaccine in Indian children in the second year of life. Vaccine. 2014 Aug 11;32 Suppl 1:A110-6. doi: 10.1016/j.vaccine.2014.04.079. PMID 25091663
- [Derived] Bhandari N, Rongsen-Chandola T, Bavdekar A, John J, Antony K, Taneja S, Goyal N, Kawade A, Kang G, Rathore SS, Juvekar S, Muliyil J, Arya A, Shaikh H, Abraham V, Vrati S, Proschan M, Kohberger R, Thiry G, Glass R, Greenberg HB, Curlin G, Mohan K, Harshavardhan GV, Prasad S, Rao TS, Boslego J, Bhan MK; India Rotavirus Vaccine Group. Efficacy of a monovalent human-bovine (116E) rotavirus vaccine in Indian infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2014 Jun 21;383(9935):2136-43. doi: 10.1016/S0140-6736(13)62630-6. Epub 2014 Mar 12. PMID 24629994